CLINICAL TRIAL: NCT01296763
Title: A Randomized Multi-center Phase I/II Trial of ICM (Irinotecan, Cisplatin, Mitomycin C) With or Without AZD2281 (Olaparib) in Patients With Advanced Pancreatic Cancer
Brief Title: Trial of ICM With or Without AZD2281 (Olaparib) in Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1070; RC2CA148346-01 (NIH); NA_00032826 (Other: JHMIRB)
Record Dates: First submitted 2011-01-21; First posted 2011-02-15 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-02

CONDITIONS: Pancreatic Cancer
Keywords: Irinotecan; Cisplatin; Carboplatin; Mitomycin-C; Olaparib; AZD2281
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Irinotecan; Cisplatin; olaparib; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan, Cisplatin, Olaparib, then add Mitomycin-C (Experimental): A 3+3 dose escalation design will be used starting with dose 1. The maximally tolerated dose is defined as the highest dose for which at most 1 out of 6 patients experiences a DLT. We will use 3 patients per dose cohort. If 0 of 3 patients have a DLT (see section 5a) then the escalation will be continued at the next dose level. If 1 of 3 patients have a DLT then three more patients will be enrolled at this dose. If 1 of 6 patients has a DLT then the dose escalation will continue. If 2 or more of the first 3 patients, or >2 of 6 patients treated have a DLT at the dose level, we will reduce the dose to the previous dose level of Olaparib for the phase 2 and then test Mitomycin C (phase 1 dose 5). If DLTs are observed at our dose 1 regimen, we will reduce the duration of Olaparib from day 1 and day 8 to just day 1 (dose level -1) and we will not test Mitomycin C in the trial.
  Interventions: Drug: Irinotecan; Drug: Cisplatin; Drug: Olaparib (for levels 1 and 5); Drug: Olaparib (for dose level 2); Drug: Mitomycin-C

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 70 mg/m2 IV, Days 1 and 8
Drug: Cisplatin — Cisplatin 25 mg/m2 IV, Days 1 and 8
Drug: Olaparib (for levels 1 and 5) — Olaparib 100 mg bid oral, Days 1 and 8
Drug: Olaparib (for dose level 2) — Olaparib 100mg bid oral, Day 1-3, Day 8-10
Drug: Mitomycin-C — Mitomycin 5 mg/m2 IV, Day 1

SUMMARY:
Patients whose pancreatic cancers have defects in the BRCA/Fanconi DNA repair pathway or other defects in homologous repair will have cancers that respond to olaparib when given in combination with the DNA damaging agents, irinotecan, cisplatin, mitomycin C (ICM).

DETAILED DESCRIPTION:
The trial is designed to evaluate the role of Parp inhibitor based therapy, combining the most well studied and potent Parp inhibitor currently available with a low-dose combination of DNA damaging agents to optimize the effects of Parp inhibition. To ensure optimal response rates in the trial, to enrich our population for patients likely to achieve the best clinical response to Parp inhibitor based therapy, we will recruit and enroll patients with known BRCA mutations, patients of Jewish ancestry, patients with familial pancreatic cancer, as well as with sporadic pancreatic cancer. We will test patients and their cancers for other inherited or acquired defects in homologous DNA repair. For the phase 1 study, we will enroll up to 30 patients. For the phase 2 component of the study, 100 patients with locally, advanced, unresectable or metastatic pancreatic cancer will be enrolled. An initial phase I analysis will be performed to test the safety of the ICM with Olaparib regimen at the doses we predict will be effective for the phase 2 and ensure that these doses are below the maximum tolerated dose. For this phase 1 we will use a standard 3+3 design and will test the following dose regimens in a 28 day cycle:

Dose level 1: Cisplatin/Irinotecan i.v.(day 1, 8) and Olaparib (100 mg bid p.o., Day 1 & Day 8) Dose level 2: Cisplatin/Irinotecan i.v.(day 1, 8) and Olaparib 100 bid p.o. day 1-3, day 8-10 (if this dose is not tolerated, go to Dose 5: Mitomycin + Olaparib Dose level 1) Dose level 3: Cisplatin/Irinotecan i.v.(day 1, 8) and Olaparib 200 bid p.o.day 1-3, day 8-10 (if this dose is not tolerated, go to Dose 5: Mitomycin + Olaparib Dose level 2) Dose level 4: Cisplatin/Irinotecan i.v.(day 1, 8) and Olaparib 200 bid p.o. day 1-12 (if this dose is not tolerated, go to Dose 5: Mitomycin + Olaparib Dose level 3)) Dose level 5: Cisplatin/Irinotecan i.v.(day 1, 8), Mitomycin Day 1 (5 mg/m2 IV), along with the established tolerated dose level of Olaparib.

Other intermediate dose schedules of Olaparib may be considered to achieve the most optimal tolerable regimen" If there are DLTs at Dose 1, we will reduce the duration of Olaparib

Note: The Principal Investigator and Astrazeneca decided not to move forward with the Phase II part of the study. Therefore the arms of Irinotecan, Cisplatin, Mitomycin C with Olaparib versus Irinotecan, Cisplatin, Mitomycin C without Olaparib will not be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Histologic or cytologic confirmation of exocrine pancreatic adenocarcinoma.
3. Locally advanced, inoperable (due to venous or arterial encasement ≥ 180° of the vessel), and/or metastatic disease by imaging (CT, MRI, or EUS). Acquisition of tissue rather than cytology is encouraged if the patient gives informed consent.
4. Measurable disease according to RECIST 1.1 criteria
5. Prior neoadjuvant or adjuvant therapy is acceptable, as long as no more than one drug of the ICM regimen was used.
6. No prior chemotherapy for advanced pancreatic cancer with Olaparib is permitted. Gemzar, Tarceva, and 5-FU or Xeloda, Oxaliplatin Taxotere, and FOLFIRINOX are permitted.
7. Three weeks since last surgery or chemotherapy mentioned in #5 above or investigational therapies. Four weeks since radiation.
8. No prior PARP inhibitors of any type
9. ECOG status < 3
10. Life expectancy > 3 months
11. Patients must have normal organ and bone marrow function
12. Age >=18.
13. Patient is willing and able to comply with the protocol for the duration of the study including treatment, scheduled visits, and examinations.
14. Evidence of non-childbearing status for women of childbearing potential, or postmenopausal status: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1

    For inclusion in genetic research, patients must fulfill the following criterion:
15. Provision of informed consent for genetic research. If a patient declines to participate in the genetic research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study.

Exclusion Criteria:

1. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer or curatively treated in-situ solid tumors with no evidence of disease for ≥ 5 years.
2. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), less than 3 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates for bone metastases before and during the study as long as these were started at least 4 weeks prior to treatment.
3. For patients who have locally advanced pancreatic cancer only, if they have received therapeutic doses of radiation therapy to their pancreatic bed (~50 Gy) for treatment of their locally advanced pancreatic cancer
4. Patients having already had prior chemotherapy for more than 12 months for their advanced pancreatic cancer (not including adjuvant/neoadjuvant)
5. Patients receiving the following classes of inhibitors of CYP3A4 (see Section for guidelines and wash out periods).
6. Current use of azole antifungals, macrolide antibiotics, or protease inhibitors
7. Unresolved toxicities (>CTCAE 4.0 grade 2) caused by previous cancer therapy.
8. Patients with known brain metastases. A scan to confirm the absence of brain metastases is not required unless the initial examination reveals CNS signs of disease.
9. Major surgery less than 3 weeks prior to starting study treatment and patients must have recovered from any effects of any major surgery.
10. Patients considered a poor medical risk due to serious, uncontrolled medical disorders, non-malignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
11. Patients unable to swallow oral medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
12. Breast feeding and/or pregnant women.
13. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
14. Patients with known active hepatic disease (i.e., Hepatitis B or C). Patients with a known hypersensitivity to Olaparib or any of the excipients of the product or history of severe allergic reactions to platinums or chemotherapy.
15. Grade 2 neuropathy at entry from any etiology, including diabetes (in view of Cisplatin).
16. Prior episodes of recurrent deep vein thrombosis or Trousseau's Syndrome unless the patient is successfully anticoagulated. If a patient has had a history of clotting or is suspected to have Trousseau's syndrome and is not anticoagulated, a D-Dimer level will be checked. If it is > 3 x ULN, patients will be expected to be anticoagulated with low molecular weight heparinoids (i.e. Lovonox).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goggins, MD, Principal Investigator — Sol Goldman Pancreatic Cancer Research Center, JHMI
Locations (2):
- United States (2):
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Columbia University Medical Center, New York, New York

REFERENCES:
- [Derived] Yarchoan M, Myzak MC, Johnson BA 3rd, De Jesus-Acosta A, Le DT, Jaffee EM, Azad NS, Donehower RC, Zheng L, Oberstein PE, Fine RL, Laheru DA, Goggins M. Olaparib in combination with irinotecan, cisplatin, and mitomycin C in patients with advanced pancreatic cancer. Oncotarget. 2017 Jul 4;8(27):44073-44081. doi: 10.18632/oncotarget.17237. PMID 28454122

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 1. Irinotecan 70 mg/m2 IV, Days 1 and 8
  2. Cisplatin 25 mg/m2 IV, Days 1 and 8
  3. Olaparib 100 mg bid oral, Days 1 and 8
- Dose Level 2: 1. Irinotecan 70 mg/m2 IV, Days 1 and 8
  2. Cisplatin 25 mg/m2 IV, Days 1 and 8
  3. Olaparib 100mg bid oral, Day 1-3, Day 8-10
- Dose Level 5: 1. Irinotecan 70 mg/m2 IV, Days 1 and 8
  2. Cisplatin 25 mg/m2 IV, Days 1 and 8
  3. Mitomycin 5 mg/m2 IV, Day 1
  4. Olaparib 100 mg bid oral, Days 1 and 8
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 5
Started | 7 | 5 | 6
Completed | 7 | 5 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subject with advanced pancreatic cancer
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 5 | Total
Number analyzed (Participants) | 7 | 5 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 5 | 15
  >=65 years | 0 | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 59.28 [47.31 to 65.81] | 59.08 [33.09 to 72.9] | 51.98 [38.73 to 76.48] | 56.79 [33.09 to 76.48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 9
  Male | 4 | 1 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 5 | 5 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 7 | 5 | 5 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity to Determine the Maximum Tolerated Dose (MTD)
Description: 1.Phase I - Assess the safety and toxicities of IC with Olaparib escalating to ICM with Olaparib in patients with locally advanced and metastatic pancreatic cancer and determine the phase 2 dose. The number of subjects who experienced a dose limiting toxicity was assessed.Dose-limiting toxicity (DLT) is defined as any of the following study drug-related events experienced during Cycle 1:
  Thrombocytopenia with platelets <25,000 x106/l > 7 days. Grade 4 neutropenia lasting ≥7 days. Grade 3 or 4 febrile neutropenia. Grade 3 or greater non-haematological toxicities; excluding grade 3 diarrhoea, nausea or vomiting despite adequate treatment and grade 3 fatigue, lethargy and GGT elevation.
  Delay of >2 weeks for next scheduled IC/ICM for reasons of toxicity.
Time Frame: 2 years
Population: Number of subjects who experienced a dose limiting toxicity, as defined in the protocol.
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 5
Number analyzed (Participants) | 7 | 5 | 6
participants | 0 | 2 | 2

2. Secondary Outcome: Number of Years From Cycle 1, Day 1 On-Study to Date of Death
Description: The overall survival of subjects with locally advanced and/or metastatic pancreatic cancer treated with Irinotecan, Cisplatin, Olaparib, with escalation to the addition of Mitomycin-C. Survival from cycle 1, day 1 on-study to date of death was assessed.
Time Frame: 5 years
Measure: Mean (Full Range); unit: years (survival) from C1D1 to death
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 5
Number analyzed (Participants) | 7 | 5 | 6
years (survival) from C1D1 to death | 1.43 [0.06 to 4.46] | 0.44 [0.08 to 1.03] | 0.60 [0.13 to 1.58]

ADVERSE EVENTS:
Time Frame: up to 30 days after end of study visit.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 5
Serious Adverse Events (participants affected / at risk) | 5/7 | 4/5 | 4/6
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=7) | Dose Level 2 (N=5) | Dose Level 5 (N=6)
Myelodysplastic syndrome (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
hemorrhagic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
prolapsed colostomy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
atrial fibrilation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
right fronto-temporal subdural hematoma (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=7) | Dose Level 2 (N=5) | Dose Level 5 (N=6)
abdominal ascites (Gastrointestinal disorders) | 1 | 0 | 1
abdominal cramps (Gastrointestinal disorders) | 0 | 1 | 1
abdominal distention (Gastrointestinal disorders) | 1 | 0 | 1
abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
alk phos increased (Investigations) | 3 | 2 | 3
alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
ALT increased (Investigations) | 3 | 2 | 3
anemia (Blood and lymphatic system disorders) | 7 | 3 | 5
anorexia (Metabolism and nutrition disorders) | 4 | 0 | 3
anticipatory nausea (Gastrointestinal disorders) | 1 | 0 | 0
anxiety (Psychiatric disorders) | 1 | 0 | 0
AST increased (Investigations) | 2 | 2 | 3
asthenia (General disorders) | 0 | 0 | 2
atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
bilirubin increased (Investigations) | 1 | 2 | 0
bloody stools (Gastrointestinal disorders) | 1 | 0 | 0
blurry vision (Eye disorders) | 0 | 0 | 1
dry eyes (Eye disorders) | 0 | 0 | 1
bruising around port (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
chest pain (General disorders) | 1 | 0 | 1
chills (General disorders) | 3 | 0 | 0
clogged ear (Ear and labyrinth disorders) | 0 | 0 | 1
confusion (Psychiatric disorders) | 0 | 0 | 1
congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
constipation (Gastrointestinal disorders) | 1 | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
creatinine increased (Investigations) | 3 | 2 | 2
dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2
depression (Psychiatric disorders) | 0 | 1 | 0
diarrhea (Gastrointestinal disorders) | 3 | 3 | 2
difficulty swallowing (Gastrointestinal disorders) | 1 | 0 | 1
difficulty urinating (Renal and urinary disorders) | 1 | 0 | 0
dizziness (Nervous system disorders) | 0 | 1 | 1
dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
dysgeusia (Nervous system disorders) | 0 | 0 | 2
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
edema (General disorders) | 2 | 0 | 1
fatigue (General disorders) | 5 | 2 | 4
fever (General disorders) | 3 | 2 | 1
flushing (Vascular disorders) | 0 | 0 | 2
gastritis (Gastrointestinal disorders) | 1 | 0 | 0
gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0
green mucous (nose) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
head cold with nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
headache (Nervous system disorders) | 0 | 1 | 1
heart palpitations (Cardiac disorders) | 1 | 0 | 0
heartburn (Gastrointestinal disorders) | 1 | 0 | 2
hematemesis (Gastrointestinal disorders) | 1 | 0 | 0
hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
hoarseness (int) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
hyperglycemia (Metabolism and nutrition disorders) | 5 | 4 | 4
hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
hyperphosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 0
hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 3 | 2
hypocalcemia (Metabolism and nutrition disorders) | 3 | 3 | 3
hypoglycemia (low) (Metabolism and nutrition disorders) | 0 | 1 | 0
hypokalemia (Metabolism and nutrition disorders) | 3 | 3 | 4
hypomagnesemia (Metabolism and nutrition disorders) | 2 | 3 | 1
hyponatremia (Metabolism and nutrition disorders) | 2 | 2 | 3
hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 0
hypotension (Vascular disorders) | 1 | 1 | 0
incontinent of stool (Gastrointestinal disorders) | 1 | 1 | 0
increased urination (including at night) (intermittent) (Renal and urinary disorders) | 1 | 0 | 0
infection (cold symptoms) (Infections and infestations) | 0 | 0 | 1
insomnia (Psychiatric disorders) | 1 | 0 | 1
itching skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
jaundice (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
knee pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
lymphocytes decreased (Investigations) | 7 | 3 | 6
memory impairment (intermittent) (Nervous system disorders) | 0 | 0 | 1
mucositis (Gastrointestinal disorders) | 0 | 0 | 1
muscle aches (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
nausea (Gastrointestinal disorders) | 4 | 3 | 5
neuropathies (Nervous system disorders) | 1 | 0 | 2
neutrophils decreased (Investigations) | 7 | 3 | 6
night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
nocturia (Renal and urinary disorders) | 1 | 0 | 0
nose bleed (epistaxis) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
otitis media (Ear and labyrinth disorders) | 0 | 1 | 0
pain in groin (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
platelets decreased (Investigations) | 6 | 4 | 6
post nasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
pressure in sternal area (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
PT increased (Investigations) | 0 | 3 | 2
PTT increased (Investigations) | 3 | 2 | 3
rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
rash (left ear) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
rectal bleeding (Gastrointestinal disorders) | 1 | 0 | 0
skin redness, swelling, right arm (shoulder to elbow) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
runny nose (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
sepsis (Infections and infestations) | 1 | 1 | 0
sore throat (Infections and infestations) | 0 | 1 | 1
stiffness in abdomen (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
stomach pain (Gastrointestinal disorders) | 0 | 0 | 1
stomach virus recovery (Gastrointestinal disorders) | 1 | 0 | 0
stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
stool leakage (Gastrointestinal disorders) | 1 | 0 | 0
stuffy nose (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
syncope (Nervous system disorders) | 2 | 0 | 0
tearing (watery eyes) (Eye disorders) | 0 | 0 | 2
tremors (Nervous system disorders) | 1 | 0 | 0
upper respiratory infection (Infections and infestations) | 1 | 0 | 0
vomiting (Gastrointestinal disorders) | 3 | 3 | 5
WBC decreased (Investigations) | 7 | 5 | 6
weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
weight loss (Investigations) | 2 | 0 | 1

LIMITATIONS AND CAVEATS:
The P.I. and Astrazeneca decided not to move forward with the Phase II part of the study. Therefore the arms of Irinotecan, Cisplatin, Mitomycin C with Olaparib versus Irinotecan, Cisplatin, Mitomycin C without Olaparib will not be compared.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes